CLINICAL TRIAL: NCT00263302
Title: Diuretic Efficacy of Dexamethasone in Congestive Heart Failure Patients
Brief Title: Diuretic Efficacy of Dexamethasone in Heart Failure
Status: Suspended | Phase: Phase 1 | Type: Interventional
Sponsor: Hebei Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0512-e
Record Dates: First submitted 2005-12-07; First posted 2005-12-08 (Estimated); Last update posted 2008-07-04 (Estimated); Status verified 2005-01

CONDITIONS: Heart Failure, Congestive
Keywords: dexamethasone, diuretic, congestive heart failure
MeSH Terms: conditions — Heart Failure | interventions — Dexamethasone

INTERVENTIONS:
Drug: dexamethasone

SUMMARY:
The purpose of this study is to determine whether glucocorticoids have potent diuretic effects in patients with congestive heart failure.

DETAILED DESCRIPTION:
Glucocorticoids are known to have pronounced physiological effects in the kidney. Conventional teaching dictates that it should be used with caution in patients with congestive heart failure due to its fluid and sodium retention effects. Surprisingly, despite the widespread prevalence of this belief within the medical community, there are few data to support it. In fact, several small animal studies have documented its striking diuretic effects due to increased renal plasma flow and glomerular filtration rate without changes in the glomerular filtration fraction. We design this study to determine whether glucocorticoids have a potent diuretic effect in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Congestive heart failure patients due to any cause
* Patients with normal cortical function
* Congestive heart failure patients who are on diuretic therapy
* Clinically stable and body weight maintained the same for at least 3 days without signs of fluid retention

Exclusion Criteria:

* Patient refusal
* Signs of infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2006-03; Study Completion 2006-12

PRIMARY OUTCOMES:
urine volume
urine electrolyte excretion (urine sodium, urine potassium, urine chloride), and urine creatinine.
serum electrolyte (serum sodium, serum potassium, serum chloride), serum creatinine, serum urea, serum uric Acid.
fractional sodium excretion
glomerular filtration rate (calculated by Cockroft and Gault formula).

CONTACTS AND LOCATIONS:
Overall Officials: Kunshen Liu, M.D., Study Chair — Hebei Medical University
Locations (2):
- China (2):
  - Kunshen Liu, Shijiazhuang, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei